CLINICAL TRIAL: NCT03322761
Title: Exercise as a Supplemental Treatment Strategy Early in the Disease Course of Multiple Sclerosis
Brief Title: Early Exercise Efforts in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Morten_Riemenschneider_PhD
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Exercise; Disease-modifying treatment; Early treatment
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systematic exercise training (Experimental): Two weekly supervised aerobic exercise trainings for 48 weeks. The training will be planned by exercise physiologists, and performed in a progressive manner.
  Interventions: Combination Product: Systematic exercise training
- Educational program (Active Comparator): Educational program on physical activity and health, consisting of four educational sessions in the intervention period.
  Interventions: Behavioral: Educational program
- Standard treatment alone (No Intervention): Data from The Danish MS Registry will serve as control-data for standard treatment alone.

INTERVENTIONS:
Combination Product: Systematic exercise training — Combination of standard medical treatment and systematic early exercise training in persons with MS.
  Arms: Systematic exercise training
Behavioral: Educational program — Informations regarding health benefits of physical activity and exercise.
  Arms: Educational program

SUMMARY:
This study seeks to investigate whether early exercise efforts can expand the use of exercise in Multiple sclerosis (MS), from symptom treatment only, to early supplementary disease-modifying treatment.

The study will be conducted in a randomized and controlled manner, with single blinding. Participants will be allocated to either a systematic aerobic exercise intervention or an educational programme on exercise and physical activity. Both interventions will last 1 year, and involve a 1 year follow-up period.

It is hypothesized that early exercise efforts can modify the disease activity and disability progression.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an autoimmune and neurodegenerative disease in the central nervous system (CNS), characterized by a complex pathogenesis and heterogeneous symptoms. The histopathological hallmark of the disease is sclerotic lesions. These inflammatory lesions manifests as disabling relapses, and the number of relapses in the first few years after disease onset is associated with progression of disability, with a higher number of relapses leading to a more rapid progression. In addition, diffuse neurodegeneration seems to occur early in the disease, and even though it is not always clinically evident it is associated with disease progression. A reduction in relapse rate and neurodegeneration early in the MS disease course may slow the progression of disabilities and can possibly reduce overall disease burden. For the individual person with MS (pwMS) a reduction in overall disease burden will often improve quality of life, and since MS is a lifelong disease this is of great interest. Preventing disability in pwMS is also highly relevant in a societal perspective, as it lowers the large costs associated with increased disability. As a consequence, the importance of early treatment have been emphasized.

Treatment of MS have seen great advances in the recent years, resulting in an increasing number of available disease-modifying treatments (DMT). Despite the fact that the current DMTs favourable alter a number of clinical outcomes and the course of the disease, it is still a serious and deteriorating condition with significant disease activity, impaired neurological functions and thus progression of disabilities. New and supplemental treatment strategies are therefore still warranted, and exercise have gained attention as a safe and tolerable rehabilitation strategy. Recently, exercise furthermore have gained substantial attention, as the first indications of neuroprotective and disease-modifying effects of exercise has been published. However, despite the focus on early treatment in medical DMTs no studies have investigated the effects of exercise as a supplemental treatment strategy early in the disease course of MS.

Consequently, the purpose of this study is to investigate the effects of early exercise efforts on disease activity and disability progression. In a sub-group the effects will furthermore be investigated on brain volume, specific brain regions, and inflammation.

It is hypothesized that early exercise efforts can modify the disease activity and disability progression, by reducing the relapse rate, the progression of Multiple Sclerosis Functional Composite (MSFC) and Expanded Disability Status Scale (EDSS) scores. The rate of brain atrophy and the lesion load, obtained by MRI scans, is also hypothesized to be reduced. This is expected to be due to an exercise-induced reduction in inflammation.

The study will be a randomised and controlled study with randomisation to either an systematic aerobic exercise intervention or an educational programme on exercise and physical activity. Both interventions are in addition to standard treatment, and will last 1 year. The exercise intervention will consist of 2 supervised exercise sessions per week in the complete duration of the study, while the standard treatment plus exercise education program will consist of 4 educational sessions on the health benefits associated with exercise and physical activity held every third month throughout the intervention period. The training in the exercise group will be aerobic exercise (running, cycling, rowing or on a cross-trainer) planned by exercise physiologists and performed in a progressive manner. To allow handling of a large number of participants, who is also geographically spread, the exercise intervention will be locally anchored, but at the same time supervised by student employees from Section for Sports Science and controlled by internet- and telephonic communication. In addition to the two intervention groups, data from The Danish MS registry will serve as population based standard treatment control data. All groups will be followed up 1 year after cessation of the interventions.

To set the estimated number of participants a two-sample two-sided power calculation has been conducted. The basis for this calculation is an report from Tallner et al. who have shown a difference in relapse rate during a two-year period (equal to our 1 year intervention, and 1 year follow-up) of 0.65 relapses between physically active and physically inactive MS patients (active: 0.95 +/- 0.97 relapses in 2 years ; inactive: 1.60 +/- 1.64 relapses in 2 years). 83 patients with MS should be enrolled in each intervention group (a 20% drop-out rate has been included). Newly published data on the brain atrophy in percentage of total brain volume after 24 weeks of resistance training have been the basis for a similar calculation of the number of participants in the sub-group, from whom MRI-scans and blood samples will be obtained. 41 participants from each intervention group should form this sub-group.

MS is a complex disease with heterogenous symptoms, and by combining the disciplines of exercise physiology, neurology and radiology this study can be the first long-term and large-scale exercise study to investigate the possible neuroprotective and disease-modifying effects of exercise when initiated early in the disease course of MS. Consequently, this project has the potential to change present clinical practice and generate further attention to exercise, not only as symptom treatment, but also as an supplemental disease-modifying treatment strategy early in the course of MS.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Definite diagnosis with Relapsing remitting multiple sclerosis (RRMS)
* No more than 2 years since diagnosis
* Expectedly able to carry out high intensity aerobic training
* Able to transport themselves to and from training sessions

Exclusion Criteria:

* Pregnancy
* Dementia, alcohol abuse, or pacemaker
* Metallic implants, hindering MRI-scans
* Comorbidities hindering participation in high intensity aerobic training

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Annual Relapse Rate (ARR) | ARR, 1 year intervention; 1 year follow up.
  Number of relapses, registered and validated by neurologist, on annual basis
Percentage brain volume change | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Brain atrophy will be measured from MRI-scans

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Composite score from Timed 25-Feet Walk Test (T25FWT), 9-Hole Peg Test (9HPT), Paced Auditory Serial Addition Test (PASAT)
Expanded Disability Status Scale (EDSS) score | Baseline, after 1 year intervention, and again at 1 year follow up.
  Disability status score assessed and registered by neurologist. The scale ranges from 0-10 in 0.5 unit increments representing higher levels of disability.

OTHER OUTCOMES:
Functional capacity, Six-minute walk test (6MWT) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Distance covered during a six-minute maximal walking test
Functional capacity, Six-spot-step-test (SSST) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  SSSt is a measure of walking ability, balance and coordination. Measured as the time to complete the six-spot course.
Functional capacity, Accelerometry | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Measurement of level of physical activity by wearing a accelerometer for 7 days at each timepoint. Measured in counts/min.
Aerobic capacity | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Maximal oxygen uptake test on bike ergometer, measured by indirect calorimetry.
Cognition, Symbol Digit Modality Test (SDMT) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Assessment of cognitive function (processing speed), with a higher number of correct answers in the test representing better cognitive function.
Cognition, Paced Auditory Serial Addition Test (PASAT) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Assessment of cognitive function (processing speed and memory), with a higher number of correct answers in the test representing better cognitive function.
Cognition, Selective Reminding Test (SRT) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Assessment of cognitive function (memory), with a higher number of correct answers in the test representing better cognitive function.
Short Form Health Survey 36 (SF-36) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Questionnaire assessing health status. The SF-36 consists of eight subscales, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Multiple Sclerosis Impact Scale 29 (MSIS-29) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Questionnaire assessing the impact of the disease. 20 questions measure the physical impact, and 9 questions measure the psychological impact. Each question is scored from 1-5. A greater score is equal to a larger impact.
Multiple Sclerosis Walking Scale 12 (MSWS-12) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Questionnaire assessing the impact of the disease on walking. Each question is scored from 1-5 and then summed and transformed to a 0-100 scale. Higher scores indicate a greater impact on walking.
Modified Fatigue Impact Scale (MFIS) | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Questionnaire assessing the effects of fatigue on physical, cognitive and psychosocial functioning. The score of the MFIS is the sum of the scores for the 21 items. A higher score represents a higher impact of fatigue, in general or in relation to one of the above mentioned areas.
Number of lesions | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Number of lesions, measured by MRI-scanning.
Lesion load | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Volume of lesions, measured by MRI-scanning.
Kurtosis | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  MRI-measure of microstructural changes in the brain
Inflammation | Baseline, 24 weeks, after 1 year intervention, and again at 1 year follow up.
  Blood samples will be analyzed for key inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Morten Riemenschneider, MSc, Principal Investigator — Section for Sport Science, Department of Public Health, Aarhus University
Locations (1):
- Section for Sport Science, Department of Public Health, University of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data will be stored in The Danish National Archives after completion of the project, and data can be accessed through request to The Danish National Archives.
Time Frame: The data will become available after completion of the project, expectedly January 2021. The Danish National Archives stores data without a time frame (forever).
Access Criteria: Sharing of data can happen upon request to The Danish National Archives.

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Ziemssen T, De Stefano N, Sormani MP, Van Wijmeersch B, Wiendl H, Kieseier BC. Optimizing therapy early in multiple sclerosis: An evidence-based view. Mult Scler Relat Disord. 2015 Sep;4(5):460-469. doi: 10.1016/j.msard.2015.07.007. Epub 2015 Jul 17. PMID 26346796
- [Background] Patwardhan MB, Matchar DB, Samsa GP, McCrory DC, Williams RG, Li TT. Cost of multiple sclerosis by level of disability: a review of literature. Mult Scler. 2005 Apr;11(2):232-9. doi: 10.1191/1352458505ms1137oa. PMID 15794399
- [Background] Wingerchuk DM, Carter JL. Multiple sclerosis: current and emerging disease-modifying therapies and treatment strategies. Mayo Clin Proc. 2014 Feb;89(2):225-40. doi: 10.1016/j.mayocp.2013.11.002. PMID 24485135
- [Background] Elovaara I. Early treatment in multiple sclerosis. J Neurol Sci. 2011 Dec;311 Suppl 1:S24-8. doi: 10.1016/S0022-510X(11)70005-3. PMID 22206762
- [Background] Dalgas U, Stenager E, Ingemann-Hansen T. Multiple sclerosis and physical exercise: recommendations for the application of resistance-, endurance- and combined training. Mult Scler. 2008 Jan;14(1):35-53. doi: 10.1177/1352458507079445. Epub 2007 Sep 19. PMID 17881393
- [Background] Kjolhede T, Siemonsen S, Wenzel D, Stellmann JP, Ringgaard S, Pedersen BG, Stenager E, Petersen T, Vissing K, Heesen C, Dalgas U. Can resistance training impact MRI outcomes in relapsing-remitting multiple sclerosis? Mult Scler. 2018 Sep;24(10):1356-1365. doi: 10.1177/1352458517722645. Epub 2017 Jul 28. PMID 28752800
- [Derived] Kupjetz M, Langeskov-Christensen M, Riemenschneider M, Inerle S, Ligges U, Gaemelke T, Patt N, Bansi J, Gonzenbach RR, Reuter M, Rosenberger F, Meyer T, McCann A, Ueland PM, Eskildsen SF, Nygaard MKE, Joisten N, Hvid L, Dalgas U, Zimmer P. Persons With Multiple Sclerosis Reveal Distinct Kynurenine Pathway Metabolite Patterns: A Multinational Cross-Sectional Study. Neurol Neuroimmunol Neuroinflamm. 2025 Nov;12(6):e200461. doi: 10.1212/NXI.0000000000200461. Epub 2025 Sep 18. PMID 40966534
- [Derived] Riemenschneider M, Hvid LG, Petersen T, Stenager E, Dalgas U. Exercise Therapy in Early Multiple Sclerosis Improves Physical Function But Not Cognition: Secondary Analyses From a Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 May;37(5):288-297. doi: 10.1177/15459683231159659. Epub 2023 Mar 10. PMID 36905131
- [Derived] Riemenschneider M, Hvid LG, Ringgaard S, Nygaard MKE, Eskildsen SF, Petersen T, Stenager E, Dalgas U. Study protocol: randomised controlled trial evaluating exercise therapy as a supplemental treatment strategy in early multiple sclerosis: the Early Multiple Sclerosis Exercise Study (EMSES). BMJ Open. 2021 Jan 12;11(1):e043699. doi: 10.1136/bmjopen-2020-043699. PMID 33436475